CLINICAL TRIAL: NCT04584502
Title: Mindful Moms in Recovery: Yoga-based Mindfulness Relapse Prevention for Pregnant Women With Opioid Use Disorder
Brief Title: Mindful Moms in Recovery
Acronym: MMORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sarah E. Lord, Director, Dissemination and Implementation Science Core, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00031364; R33AT010117 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Opioid-use Disorder
Keywords: Pregnancy; Mindfulness; Yoga; Substance Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Intervention as adjunct to usual care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study will be blind to the Principal Investigators, the statistician, and to those on the team responsible for participant data collection. The study team will work to try to blind clinicians delivering treatment as usual to participant assignment but there is a chance that patients will reveal their condition to clinicians despite our best efforts. To achieve blindness, treatment assignment will done by the Project Manager, who will not be directly involved in evaluation data collection. Data collection will be conducted by the study Research Assistant who will be blinded to participant treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention as adjunct to Treatment as Usual (Experimental): Participants will attend via Zoom an 8-session group-based yoga-mindfulness intervention offered over the course of approximately 10 consecutive weeks. Participants will also be asked to use a mobile companion app once a week during the intervention period. All intervention participants also receive treatment as usual for OUD at the partner practice, which includes medication for OUD, individual and/or group counseling, and case management.
  Interventions: Behavioral: Mindful Moms Yoga Mindfulness Intervention
- Treatment as Usual (No Intervention): Participants receive treatment as usual for OUD at the partner practice, which includes medication for OUD, individual and/or group counseling, and case management.

INTERVENTIONS:
Behavioral: Mindful Moms Yoga Mindfulness Intervention — MMORE is an 8-session yoga-mindfulness intervention protocol, offered via Zoom over the course of 10 consecutive weeks at the partner maternity care practice or a nearby location. Each session will last approximately 60 minutes (8 - 10 participants per group). Intervention participants will also be asked to use a mobile companion app at least once each week of the intervention period.
  Other Names: MMORE
  Arms: Intervention as adjunct to Treatment as Usual

SUMMARY:
The purpose of this study is to evaluate the initial efficacy of a yoga-mindfulness intervention to promote ongoing recovery for pregnant and parenting women with Opioid Use Disorder (OUD) receiving perinatal services and medication treatment for OUD from maternity care practices in New Hampshire.

DETAILED DESCRIPTION:
In this R33 project, the study team will conduct a randomized controlled trial to evaluate the efficacy and implementation of the Mindful Moms intervention (MMORE) with a group of pregnant women with identified OUD receiving medication treatment for OUD at partner maternity care practices. The study team will evaluate the impact of Mindful Moms as an adjunct to treatment as usual on retention in medication for opioid use disorder (MOUD) treatment, substance use, and relapse-related risks.

This study has three Specific Aims:

Aim 1: Evaluate MMORE in a randomized controlled study with pregnant women as an adjunct to MOUD treatment as usual care for impact on treatment retention, opioid abstinence, and relapse risks.

Aim 2: Examine mechanisms of effect of MMORE on outcomes.

Aim 3: Evaluate barriers and facilitators to sustainable implementation of MMORE as an adjunct to MOUD for pregnant and parenting women.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* English-speaking.
* Singleton pregnancy.
* Receiving comprehensive medication treatment for opioid use disorder as part of prenatal care at a partner maternity care practice.

Exclusion Criteria:

* Cognitive or psychiatric impairments that prohibit being able to provide informed consent.
* Any physical conditions that prohibit activity such as gentle yoga.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Lord, PhD, Principal Investigator — Geisel School of Medicine
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Significant recruitment challenges due to narrow eligibility (buprenorphine received in maternity care setting) and COVID restrictions. Recruitment ran from April 2022 to July 2023, after institutional and funder approvals were finally obtained for the revised protocol to use a virtual intervention delivery format. Recruitment occurred through partner maternity care settings primarily with flyers placed in high patient traffic areas and clinician distribution of study materials to patients.
Pre-assignment Details: One participant enrolled but could not be contacted to complete baseline assessment.
Period: Overall Study
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All of the participants that completed Baseline were randomized into the Treatment condition. One participant that completed enrollment did not complete Baseline due to loss of contact (e.g., did not respond to repeated outreach by study team).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3
Number of Participants who Self-Reported Medication Treatment for Opioid Use [Count of Participants; unit: Participants] | 3 | 0 | 3
Number of Participants Who Self-Reported Opioid and Other Substance use [Count of Participants; unit: Participants] | 3 |  | 3
Depression Symptoms [Mean (Standard Deviation); unit: units on a scale] — The Edinburgh Prenatal Depression Scale was used to assess symptoms of depression. Total scores on this 10-item measure range from 0-30, with high scores indicating higher frequency of depression symptoms. Scores >= 14 indicative of high probability of moderate-severe depression.
  units on a scale | 13.0 (1.0) |  | 13 (1.0)
Anxiety Symptoms [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder (GAD-7) screening measure was used to assess anxiety symptoms. The total score ranges from 0-21, with higher scores indicating greater frequency of anxiety symptoms. Scores >10 indicate high probability of moderate-severe anxiety.
  units on a scale | 9.7 (4.7) |  | 9.7 (4.7)
Perceived Stress [Mean (Standard Deviation); unit: units on a scale] — Measured by Perceived Stress Scale-4. The Perceived Stress Scale-4 includes 4 questions on 5-point Likert (0-4). Total scores ranging from 0 to 16 with higher scores indicating greater stress.
  units on a scale | 7.7 (.58) |  | 7.7 (.58)
Mindfulness [Mean (Standard Deviation); unit: units on a scale] — Measured by the Mindful Attention Awareness Scale, a 15-item measured on 6-point Likert scale. Higher scores associated with greater mindfulness.
  units on a scale | 3.6 (.53) |  | 3.6 (.53)
Pain [Count of Participants; unit: Participants] — no/low Pain: <5 yes/high Pain: >=5 visual analogue scale (0-10). Reported are number of participants that reported Yes/High pain symptoms.
  Participants | 0 |  | 0
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Measured by World Health Organization Quality of Life Brief instrument. Scores range from 0-100, with higher scores reflecting greater quality of life.
  units on a scale | 57.5 (5.0) |  | 57.5 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-reported Retention in Medication Treatment for Opioid Use Disorder
Description: We were not able to obtain clinical record data from partner settings due to high staff demand and considerable stress at partner settings due to the impact of COVID-19 pandemic. Data regarding retention in medication treatment was obtained via self-report in assessment surveys.
Time Frame: baseline-3-months postpartum
Population: All participants were randomly assigned to the Intervention arm.
Measure: Number; unit: participants who reported 'yes' to MOUD
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
participants who reported 'yes' to MOUD | 2 |

2. Primary Outcome: Number of Participants Who Self Reported Opioid Use
Description: We were not able to collect urine toxicology data so measured by way of self-report (frequency of use past 3 months).
  Scored as 0=No; 1=Yes
Time Frame: baseline to 3-months postpartum
Population: participants who completed 3 month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
Participants | 3 |

3. Secondary Outcome: Participant Report of Other Substance Use
Description: The Alcohol, Smoking and Substance Involvement Screening Test includes items to assess past and current substance use: tobacco, alcohol, marijuana, cocaine, heroin/fentanyl) frequency of use (past 3 months; not at all/once or twice/once a month/once or twice a month/once a week/daily or almost daily). Scored as: 0 (not at all/once or twice); 1=more than once or twice (composite of marijuana and cocaine use). Reported as # of participants that scored 1.
Time Frame: Baseline to 3-months postpartum
Population: participants that completed 3 month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
Participants | 0 |

4. Secondary Outcome: Depression Symptoms
Description: The Edinburgh Postnatal Depression Scale contains 10 questions. Total scores range from 0 to 30 with higher scores indicating greater depression symptoms.
Time Frame: Baseline to 3 months postpartum
Population: participants only randomized to intervention condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
score on a scale | 9.0 (4.6) |

5. Secondary Outcome: Anxiety Symptoms
Description: The Generalized Anxiety Disorder Scale contains 7 questions with scores ranging from 0 to 21, with higher scores indicating greater anxiety symptoms.
Time Frame: Baseline to 3-months postpartum
Population: Participants all randomized to intervention condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
score on a scale | 4.33 (4.16) |

6. Secondary Outcome: Perceived Stress
Description: The Perceived Stress Scale includes 4 questions on 5-point Likert (0-4). Total scores ranging from 0 to 16 with higher scores indicating greater stress.
Time Frame: Baseline to 3-months postpartum
Population: Participants all randomized to intervention condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
score on a scale | 5.67 (4.16) |

7. Secondary Outcome: Mindfulness
Description: The Mindful Attention Awareness Scale consists of 15 questions with scores ranging between 1 and 6 with higher mean scores indicating greater mindfulness.
Time Frame: Baseline to 3-months postpartum
Population: Participants all randomized to intervention condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
score on a scale | 4.09 (1.37) |

8. Other Pre Specified Outcome: Self-reported Quality of Life
Description: The World Health Organization Quality of Life-10 contains 10 questions to assess a quality of life profile based on four domains: physical health, psychological health, social relationships, and environment. Total score ranges from 0 to 100 where higher scores denote higher quality of life.
Time Frame: Baseline to 3-months postpartum
Population: Participants all randomized to intervention condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 3 | 0
score on a scale | 70.8 (20.2) |

ADVERSE EVENTS:
Time Frame: Baseline (pregnancy) to 3 months postpartum)(e.g., approximately 6 months).
Description: Participants all randomized Into intervention condition.
Arm/Group | Intervention as Adjunct to Treatment as Usual | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT04584502/Prot_SAP_001.pdf